CLINICAL TRIAL: NCT06216340
Title: Efficacy of Henagliflozin for Weight Loss in Obesity Without Diabetes: a Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Efficacy of Henagliflozin for Weight Loss in Obesity Without Diabetes
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Collaborators: The Second Hospital of Nanjing Medical University (Other); The First Affiliated Hospital of Soochow University (Other); Second Affiliated Hospital of Soochow University (Other); Wuxi People's Hospital (Other); Northern Jiangsu People's Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); The First People's Hospital of Lianyungang (Other); Affiliated Hospital of Jiangsu University (Other); The fourth affiliated hospital of nantong university (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-science-150
Record Dates: First submitted 2023-12-15; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Obese; Weight Loss; Pre-diabetes
Keywords: Henagliflozin; Obese; Weight loss; Glucose
MeSH Terms: conditions — Obesity; Weight Loss; Glucose Intolerance | interventions — henagliflozin

STUDY DESIGN:
Intervention Model Description: Participants are randomly divided into two groups: control group and intervention group. In control group, Placebo and diet-exercise therapy is used. In intervention group, 10mg of henagliflozin and diet-exercise therapy is used.
Who Masked: Participant, Care Provider
Masking Description: Participants and care providers are all masked. Investigators randomly cluster the participants, and the actual mask of the participant is not available to care providers and the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Placebo and diet-exercise therapy
  Interventions: Drug: Placebo
- Intervention group (Experimental): 10mg of Henagliflozin and diet-exercise therapy
  Interventions: Drug: Henagliflozin

INTERVENTIONS:
Drug: Henagliflozin — 10mg of Henagliflozin and diet-exercise therapy
  Other Names: diet-exercise therapy
  Arms: Intervention group
Drug: Placebo — Placebo and diet-exercise therapy
  Other Names: diet-exercise therapy
  Arms: Control group

SUMMARY:
This trial is conducted in China. The purpose of the 24-week trial is to investigate the efficacy of henagliflozin to induce body weight loss and the purpose of the extension is to evaluate the hypoglycemic effect of henagliflozin in obese subjects without diabetes.

Trial has the following two periods: 1) A 12-week randomized, double-blind, placebo-controlled, multi-center trial for evaluating the efficacy of henagliflozin to induce body weight loss; 2) A 12-week multicenter randomized controlled open-label trial for evaluating the hypoglycemic effect of henagliflozin followed by a 24-week extension period.

DETAILED DESCRIPTION:
Primary Hypothesis:

The 12-week henagliflozin taking could induce significantly higher weight loss in obese subjects without diabetes, compared to diet-exercise therapy.

Assessment time points:

Baseline: prior to taking henagliflozin or diet-exercise therapy V1: 4 weeks following the henagliflozin taking or diet-exercise therapy V2: 4 weeks following V1 V3: 4 weeks following V2

Specific Aims 1:

To examine and compare the weight loss, assessed by weight, waist circumference, hip circumference and BMI, after 12-week henagliflozin taking or diet-exercise therapy in obese without diabetes.

Specific Aims 2:

To examine and compare the change of glucose level after 12-week henagliflozin taking or diet-exercise therapy in obese without diabetes.

Secondary Hypothesis 1:

The 24-week henagliflozin taking could siginificantly improve the glucose control in obese subjects with pre-diabetes, compared to diet-exercise therapy.

Assessment time points:

Baseline: prior to taking henagliflozin or diet-exercise therapy V4: 12 weeks following V3

Specific Aims:

To examine and compare the change of glucose level, assessed by fasting plasma glucose (FPG), postprandial plasma glucose (PPG), HbA1c, insulin levels, after 24-week henagliflozin taking or diet-exercise therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old≤age≤65 years old, regardless of gender and race
2. Nondiabetic population: without hypoglycemic treatment, FPG<7.0 mmol/l, PPG<11.1 mmol/l, and HbA1c<6.5%
3. obesity: BMI≥28 kg/m2
4. Stable weight: weight change less than 5kg in the past 3 months
5. Ability to understand and sign the informed consent form

Exclusion Criteria:

1. Allergies to Henagliflozin or its formulations;
2. Participants have been definitely diagnosed with diabetes;
3. HbA1c≥6.5 % or FPG≥7.0 mmol/l, or PPG≥11.1 mmol/l;
4. Participants have used glucagon-like peptide-1 (GLP-1) receptor agonists, sodium glucose linked transporter-2 (SGLT-2) inhibitors, or other weight loss related drugs within the past 3 months;
5. History of bariatric surgery;
6. Untreated or uncontrolled hypothyroidism/hyperthyroidism;
7. High risk of urinary tract infection;
8. Obesity induced by other endocrinologic disorders (e.g. Cushing's Syndrome);
9. Diagnosis of congenital glucose-galactose malabsorption or familial renal glycosuria
10. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 times the upper limit of the normal range (UNL); Total bilirubin (TBIL) ≥ 2.0 times the upper limit of the normal range;
11. estimated glomerular filtration rate (eGFR)<30 mL/min/1.73 m2 or end-stage kidney disease, or requiring dialysis;
12. History of major depressive disorder or other severe psychiatric disorders, e.g. schizophrenia, bipolar disorder within the last 2 years;
13. Uncontrolled treated/untreated hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg)
14. myocardial infarction, unstable angina, revascularization surgery, or cerebrovascular diseases within the past 3 months;
15. Cancer (past or present, except basal cell skin cancer or squamous cell skin cancer) or other severe diseases, which in the investigator's opinion could interfere with the results of the trial;
16. Females of child-bearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures as required by local law or practice) within 24 months;
17. Participation in a clinical trial within the last 3 months prior to screening;
18. Previous history of gestational diabetes;
19. Previous history of eating disorders;
20. Current or history of treatment with medications that may cause significant weight gain, within 3 months prior to screening, including systemic corticosteroids (except for a short course of treatment, i.e. 7-10 days), tri-cyclic antidepressants, atypical antipsychotic and mood stabilizers (e.g. imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproic acid and its derivatives, and lithium);
21. Diet attempts using herbal supplements or over-the-counter medications within 3 months before screening
22. Any lifetime history of a suicidal attempt or a history of any suicidal behavior in the last month prior to randomization;
23. Surgery scheduled for the trial duration period, except for minor surgical procedures, at the discretion of the investigator
24. Known or suspected abuse of alcohol or narcotics
25. Subjects from the same house hold participating in the trial
26. Other situations which were inappropriate to the trial, at the discretion of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity
Enrollment: 300 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Weight change | 3 months (12 weeks)
  Proportion of weight change from baseline

SECONDARY OUTCOMES:
Proportion of ≥5% weight loss | 3 months (12 weeks)
  Proportion of patients who lost at least 5% of their body weight from baseline
Incident diabetes | 1 month (4 weeks), 2 months (8 weeks), 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), 12 months (48 weeks)
  New-onset diabetes during follow up

OTHER OUTCOMES:
Absolute weight change | 3 months (12 weeks)
  Absolute value of weight change from baseline for each group at the 3rd month
BMI change | 3 months (12 weeks)
  Change in BMI from baseline for each group at the 3rd month. BMI was defined as weight (kg) divided by height squared (m2), weight and height will be combined to report BMI in kg/m^2.
Change of waist circumference | 3 months (12 weeks)
  Change of waist circumference at the 3rd month
Change of waist-to-hip ratio | 3 months (12 weeks)
  Change of waist-to-hip ratio at the 3rd month. Waist-to-hip ratio will be defined as waist circumference (cm) to hip circumference (cm).
Change of FPG | 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), 12 months (48 weeks)
  Change of FPG from baseline
Change of PPG | 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), 12 months (48 weeks)
  Change of PPG from baseline
Changes of insulin levels | 3 months (12 weeks), 6 months (24 weeks), 12 months (48 weeks)
  Changes of fasting and oral glucose tolerance test-2h insulin level from baseline
Changes of C-peptide levels | 3 months (12 weeks), 6 months (24 weeks), 12 months (48 weeks)
  Changes of fasting and oral glucose tolerance test-2h C-peptide levels from baseline
Changes of HbA1c | 3 months (12 weeks), 6 months (24 weeks), 9 months (36 weeks), 12 months (48 weeks)
  Changes of HbA1c levels from baseline
Changes of triglyceride | 6 months (24 weeks), 12 months (48 weeks)
  Changes in triglyceride from baseline
Changes of total cholesterol | 6 months (24 weeks), 12 months (48 weeks)
  Changes in total cholesterol from baseline
Changes of LDL-c | 6 months (24 weeks), 12 months (48 weeks)
  Changes in LDL-c from baseline
Changes of HDL-c | 6 months (24 weeks), 12 months (48 weeks)
  Changes in HDL-c from baseline
Change of urinary albumin-to-creatinine ratio | 6 months (24 weeks), 12 months (48 weeks)
  Change of urinary albumin-to-creatinine ratio from baseline in each group
Changes of C-reactive protein | 6 months (24 weeks), 12 months (48 weeks)
  Changes of C-reactive protein in each group relative to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ling Yang, MD, Principal Investigator — Affiliated Hospital of Jiangsu University; Yu Liu, PHD, Principal Investigator — Nanjing Medical University; Bimin Shi, PHD, Principal Investigator — First affiliated hospital of soochow university; Ji Hu, Principal Investigator — Second Affiliated Hospital of Soochow University; Xiaowei Zhu, PHD, Principal Investigator — Wuxi People's Hospital; Zhenwen Zhang, PHD, Principal Investigator — Northern Jiangsu People's Hospital; Hongwei Ling, MD, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Ning Xu, Bachelor, Principal Investigator — The First People's Hospital of Lianyungang; Yanmei Liu, MD, Principal Investigator — YANCHENG NO.1 PEOPLE'S HOSPITAL

IPD SHARING:
Plan to Share IPD: No
The data in the current study arisen from a dataset of Department of Endocrine and Metabolic Diseases, the First People's Hospital of Changzhou, Third Affiliated Hospital of Soochow University, are not publicly available due to security consideration, but are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] WHO Guidelines on Physical Activity and Sedentary Behaviour. Geneva: World Health Organization; 2020. Available from http://www.ncbi.nlm.nih.gov/books/NBK566045/ PMID 33369898
- [Background] Wang Y, Mi J, Shan XY, Wang QJ, Ge KY. Is China facing an obesity epidemic and the consequences? The trends in obesity and chronic disease in China. Int J Obes (Lond). 2007 Jan;31(1):177-88. doi: 10.1038/sj.ijo.0803354. Epub 2006 May 2. PMID 16652128
- [Background] Wang Y, Xue H, Sun M, Zhu X, Zhao L, Yang Y. Prevention and control of obesity in China. Lancet Glob Health. 2019 Sep;7(9):e1166-e1167. doi: 10.1016/S2214-109X(19)30276-1. No abstract available. PMID 31401995
- [Background] Wang Y, Zhao L, Gao L, Pan A, Xue H. Health policy and public health implications of obesity in China. Lancet Diabetes Endocrinol. 2021 Jul;9(7):446-461. doi: 10.1016/S2213-8587(21)00118-2. Epub 2021 Jun 4. PMID 34097869
- [Background] Garvey WT, Mechanick JI, Brett EM, Garber AJ, Hurley DL, Jastreboff AM, Nadolsky K, Pessah-Pollack R, Plodkowski R; Reviewers of the AACE/ACE Obesity Clinical Practice Guidelines. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY COMPREHENSIVE CLINICAL PRACTICE GUIDELINES FOR MEDICAL CARE OF PATIENTS WITH OBESITYEXECUTIVE SUMMARYComplete Guidelines available at https://www.aace.com/publications/guidelines. Endocr Pract. 2016 Jul;22(7):842-84. doi: 10.4158/EP161356.ESGL. PMID 27472012
- [Result] American Diabetes Association Professional Practice Committee. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2022. Diabetes Care. 2022 Jan 1;45(Suppl 1):S17-S38. doi: 10.2337/dc22-S002. PMID 34964875